CLINICAL TRIAL: NCT06635707
Title: The Study on the Efficacy and Safety of Using Urapidil Alone or in Combination With Esmolol for the Treatment of Acute Hypertensive Intracerebral Hemorrhage: A Prospective, Open-label, Observational, Multicenter Research
Brief Title: Efficacy and Safety Study of Urapidil Alone or With Esmolol in Treating Acute Hypertensive Intracerebral Hemorrhage
Status: Not yet recruiting | Type: Observational
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Jianjun Wang, chief physician, Qianfoshan Hospital
Other Study IDs: YXLL-KY-2024(066)
Record Dates: First submitted 2024-09-14; First posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Hypertensive Intracerebral Hemorrhage
MeSH Terms: conditions — Intracranial Hemorrhage, Hypertensive | interventions — urapidil; esmolol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Urapidil Group: Urapidil Injection (Shijiazhuang Sipharm Co., Ltd., National Medical Products Administration Approval No. H20233626): Initially, administer a loading dose of 10mg via slow intravenous injection, observe for 5 minutes, and then adjust the infusion rate based on the patient's blood pressure, generally not exceeding 2mg/min.
  Interventions: Drug: Urapidil
- Combination Group of Urapidil and Esmolol: Urapidil Injection (Shijiazhuang Sipharm Co., Ltd., National Medical Products Administration Approval No. H20233626): Initially, administer a loading dose of 10mg via slow intravenous injection, observe for 5 minutes, and then adjust the infusion rate based on the patient's blood pressure, generally not exceeding 2mg/min.
  Esmolol Injection (Qilu Pharmaceutical Co., Ltd., National Medical Products Administration Approval No. H19991058): Administer an intravenous bolus of 1mg/kg within 30 seconds, followed by a maintenance infusion rate not exceeding 300μg/kg/min, adjusted according to blood pressure readings.
  Interventions: Drug: Urapidil and Esmolol

INTERVENTIONS:
Drug: Urapidil — 1. Control systolic blood pressure within 130-140mmHg using urapidil and maintain this level for 7 days;
  2. Reduce intracranial pressure through dehydration therapy with mannitol, positioning of the body, and other means to prevent cerebral hernia. Surgical interventions such as decompressive craniectomy may be performed if necessary;
  3. Aim for a body temperature control target of ≤37.5°C;
  4. The anticoagulation reversal target is INR < 1.5, with correction methods including the use of vitamin K, prothrombin complex concentrate (PCC), or fresh frozen plasma (FFP);
  5. The blood glucose control targets are 6.1-7.8mmol/L for non-diabetic study participants and 7.8-10.0mmol/L for diabetic study participants.
  Other Names: Ebrantil(34661-75-1)
  Groups: Urapidil Group
Drug: Urapidil and Esmolol — 1. Utilize both urapidil and esmolol to control systolic blood pressure within 130-140mmHg and maintain this level for 7 days;
  2. Reduce intracranial pressure through dehydration therapy with mannitol, strategic positioning of the body, and other measures to prevent cerebral hernia. Surgical interventions such as decompressive craniectomy may be performed if necessary;
  3. Aim for a body temperature control target of ≤37.5°C;
  4. The anticoagulation reversal target is INR < 1.5, with correction methods including the administration of vitamin K, prothrombin complex concentrate (PCC), or fresh frozen plasma (FFP);
  5. The blood glucose control targets are 6.1-7.8mmol/L for non-diabetic study participants and 7.8-10.0mmol/L for diabetic study participants.
  Other Names: 34661-75-1 and 81147-92-4
  Groups: Combination Group of Urapidil and Esmolol

SUMMARY:
The objective of this study is to investigate the efficacy and safety of urapidil monotherapy versus the combination of esmolol in treating participants with acute hypertensive intracerebral hemorrhage through a prospective, open-label, observational, multicenter clinical trial, aiming to provide guidance for clinicians in formulating rational treatment plans.

DETAILED DESCRIPTION:
Hypertensive intracerebral hemorrhage (HICH) is a prevalent and severe condition that poses significant challenges to the medical community due to its harmful nature and complexity. Over the past few decades, there has been considerable controversy surrounding blood pressure management strategies for patients with acute HICH. Both hypertension and hypotension following cerebral hemorrhage are associated with adverse outcomes. Multiple trials aimed at reducing blood pressure in patients with acute cerebral hemorrhage have been conducted, and among patients recruited within six hours of symptom onset, blood pressure reduction has been linked to decreased hematoma expansion. Current international guidelines from the European Stroke Organization, the American Heart Association (AHA)/American Stroke Association, and the Canadian Stroke Best Practice Recommendations support the prompt reduction of systolic blood pressure to 140 mmHg after symptom onset, aiming to maintain systolic blood pressure between 130 and 150 mmHg. However, for certain patients, such as those with extremely high blood pressure after ICH (systolic blood pressure >220 mmHg), a more individualized approach is necessary. Notably, patients with very high blood pressure (systolic blood pressure >220 mmHg) were not included in these trials, and reducing systolic blood pressure to 140 mmHg in this population may be harmful, associated with higher rates of neurological deterioration and adverse renal events.

Elevated blood pressure (BP) is common in patients with acute spontaneous intracerebral hemorrhage (ICH) and is closely related to hematoma growth, which is a crucial independent predictor of clinical deterioration and outcomes in ICH patients. Previous studies have shown that hematoma growth primarily occurs within the first six hours after spontaneous cerebral hemorrhage. Consequently, early blood pressure reduction may be beneficial in preventing hematoma growth. Research indicates that ICH patients who achieve target blood pressure more quickly are less likely to experience hematoma growth. Specifically, patients who reach a target systolic blood pressure (SBP) of <140 mmHg within the first hour after randomization exhibit a lower absolute hematoma growth rate. Studies have supported the benefit of shortening the time to achieve target blood pressure in ICH patients, corroborating these findings. Hematoma growth is primarily attributed to ongoing bleeding and secondary vascular rupture, occurring predominantly within the first six hours after ICH onset, particularly during the initial 2-3 hours, with a gradual decline in frequency over time.

Changes in the autonomic nervous system (ANS) have been previously observed in acute stroke patients, characterized by impaired cardiovascular regulation and altered balance between sympathetic and parasympathetic nerves. Clinically significantly, autonomic dysfunction is associated with poor prognosis, increased mortality, or sudden death after stroke. Variations in heart rate variability (HRV) and baroreceptor sensitivity (BRS) have traditionally been considered surrogate markers of cardiovascular ANS modulation. Previous studies on HRV in acute brain injury have primarily focused on ischemic cerebral infarction or traumatic brain injury (TBI). In both TBI and ischemic cerebral infarction, HRV parameters have shown independent associations with outcomes.

Urapidil (URA) is a selective α1-adrenoceptor antagonist that also acts as a central 5-HT1A receptor agonist, exerting both peripheral and central hypotensive effects. The hypotensive effect of URA is dose-dependent and may vary among individuals. URA demonstrates a self-limiting hypotensive effect, even at high doses, without causing severe hypotension. It reduces cardiac preload and afterload, decreases myocardial oxygen consumption, and increases cardiac output without causing reflex tachycardia or affecting heart rate. Additionally, URA does not increase intracranial pressure, does not impair hemodynamics in the middle cerebral artery, and is conducive to maintaining cerebral perfusion pressure. Furthermore, URA enhances renal blood flow, reduces renal vascular resistance, does not increase shunt fraction, and does not decrease arterial oxygen partial pressure.

Esmolol is an ultra-short-acting, highly selective β1-blocker that competitively antagonizes β1 receptors in myocardial cells. It exerts its pharmacological effects by blocking the activity of adrenaline and noradrenaline. At high doses, it may also block β2 receptors in airway and vascular smooth muscle. At therapeutic doses, esmolol has no intrinsic sympathomimetic activity or membrane-stabilizing effects. When administered intravenously, it takes effect within 60 seconds and its pharmacological effects disappear within 10 to 30 minutes after infusion cessation. Electrophysiological studies suggest that esmolol exhibits typical β1-blocker effects, including reduced heart rate, prolonged sinus cycle length, prolonged sinus node recovery time, prolonged AH interval and antegrade Wenckebach period, slowed conduction in atrial and ventricular myocardium and cardiac conduction system, and prolonged refractoriness. By blocking sympathetic excitation, esmolol lowers the threshold for ventricular fibrillation (VF).

Patients with acute HICH often experience increased heart rate and uncontrolled blood pressure. Previous studies have shown that the time taken to normalize blood pressure and heart rate variability are correlated with adverse outcomes in patients. The present study aims to evaluate the effectiveness of urapidil alone and in combination with esmolol in reducing blood pressure and controlling heart rate in patients with acute.

ELIGIBILITY:
Inclusion Criteria:

1. Participants in the study of acute hypertensive intracerebral hemorrhage aged between 18 and 80 years old;
2. Participants with acute intracerebral hemorrhage (basal ganglia hemorrhage < 50ml) confirmed by imaging within 6 hours of onset;
3. Participants with systolic blood pressure > 140mmHg upon admission;
4. Participants who have signed the informed consent form.

Exclusion Criteria:

1. Participants in the cerebral hemorrhage study who decline to have their disease management information collected and used and/or refuse to undergo subsequent follow-ups;
2. Participants with allergies to the medication in question;
3. Participants in the study of secondary cerebral hemorrhage resulting from tumors, vascular malformations, aneurysms, trauma, post-thrombolytic therapy, or cerebral arteriovenous thrombosis;
4. Participants undergoing anticoagulant therapy or with coagulation disorders;
5. Pregnant women;
6. Participants with multiple organ failure;
7. Participants deemed unsuitable for enrollment by the research staff due to other factors.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sample collection will be conducted for participants in the study of hypertensive intracerebral hemorrhage.
  Recruitment Locations: The First Affiliated Hospital of Shandong First Medical University (Shandong Qianfoshan Hospital), along with various other sub-centers.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Modified Rankin Scale (mRS) | Three months after the onset of the disease
  Evaluate the beneficial effect of blood pressure management with combined urapidil and esmolol on study participants by assessing the poor outcome rate, as indicated by the Modified Rankin Scale (mRS) scores (poor outcome: 4-6 points), three months after the onset of the disease.

SECONDARY OUTCOMES:
Changes in the volume of acute intracranial hematoma | First seven days of hospitalization
  Change in hematoma volume per follow-up CT
Heart rate variability | First seven days of hospitalization
  Measures of cardiac autonomic nervous system activity
Time taken for blood pressure to reach target levels after administering antihypertensive medications | First 24 hours after hospitalization
  Comparing the blood pressure-lowering ability of the two groups
Modified Rankin Scale (mRS) score | Seventh day after the onset of the disease
  Evaluate the beneficial effect of blood pressure management with combined urapidil and esmolol on study participants by assessing the poor outcome rate, as indicated by the Modified Rankin Scale (mRS) scores (poor outcome: 4-6 points)
In-hospital mortality rate | From date of randomization until the date of death from any cause, assessed up to 3 months
  Evaluation of efficacy
Mortality rate within 3 months of onset | Three months after the onset of the disease
  Response prognosis
Adverse events | During hospitalization(up to 8 weeks)
  e.g., nosocomial infections, pressure ulcers, falls, automatic discharge from hospital
Incidence of seizures | During hospitalization(up to 8 weeks)
  Cerebral hemorrhage complication rate
length of hospital stay | From date of randomization until the date of discharge from hospital for any reason, assessed up to 3 months
  Evaluation of efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Jianjun Wang, Ph.D., Study Director — Qianfoshan Hospital; Xueyan Cui, Ph.D., Study Director — Qianfoshan Hospital

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-06-24): https://cdn.clinicaltrials.gov/large-docs/07/NCT06635707/Prot_SAP_000.pdf
  • Informed Consent Form (2024-05-11): https://cdn.clinicaltrials.gov/large-docs/07/NCT06635707/ICF_001.pdf